CLINICAL TRIAL: NCT05734456
Title: Comparison Between Modified Bass and Horizontal Brushing Techniques for the Adequate Removal of Plaque in Dental Students; A Randomized Control Trial
Brief Title: Comparison Between Modified Bass and Horizontal Brushing Techniques
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CMH Lahore Medical College and Institute of Dentistry (Other)
Collaborators: Bkahtawar Amin Medical and Dental College Multan (Other); Sharif Medical Research Center (Other)
Responsible Party: Principal Investigator, Hafiz Muhammad Owais Nasim, Principal Investigator, Institute Of Dentistry, CMH LMC
Other Study IDs: CMHLahore001
Record Dates: First submitted 2023-02-03; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Tooth Plaque
Keywords: Toothbrushing technique; modified bass method; horizontal brushing technique
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to determine mean plaque scores to compare the effectiveness after using modified bass and horizontal brushing technique in undergraduate dental students. The main question[s] it aims to answer are:

* Modified bass method is less effective than the horizontal brushing technique for plaque removal in undergraduate dental students
* Modified bass method is more effective than the horizontal brushing technique for plaque in undergraduate dental students.

Participants will check plaque scores with the help of probe and disclosing agents after applying both techniques in a separate quadrant on the same subject. Researchers will compare modified bass and a horizontal brushing technique to see which one is reliable and more effective.

ELIGIBILITY:
Inclusion Criteria:

* Dental students between the ages of 19-24; irrespective of gender
* Informed consent

Exclusion Criteria:

* Students undergoing orthodontic treatment
* Students having periodontal pocket
* Students who underwent scaling less or equal to 3 months ago

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Undergraduate dental students in recognized dental colleges in Pakistan
Sampling Method: Non-Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-04-04 (Estimated); Study Completion 2023-07-04 (Estimated)

PRIMARY OUTCOMES:
Plaque Index | 24 weeks
  0-3 (0=Excellent, 3=Poor)

CONTACTS AND LOCATIONS:
Overall Officials: Mehvish Saleem, Principal Investigator — Bakhtawar Amin Medical & Dental College
Locations (1):
- Bakhtawar Amin, College of Dentistry, Multan, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT05734456/ICF_000.pdf